CLINICAL TRIAL: NCT00185172
Title: Efficacy and Safety of Olmesartan: Reduction of Blood Pressure in the Treatment of Patients Suffering From Mild to Moderate Essential Hypertension
Brief Title: Olmesartan in Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sankyo Pharma Gmbh (Industry)
Responsible Party: Senior Manager Study Coordinator, Daiichi Sankyo Europe, GmbH
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-OLM-01-00
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2008-04

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): 2 week placebo run-in
  Interventions: Other: placebo
- 2 (Experimental): Olmesartan medoxomil tablets for 8 weeks
  Interventions: Drug: olmesartan medoxomil
- 3 (Experimental): Olmesartan medoxomil tablets, or olmesartan medoxomil tablets + hydrochlorothiazide tablets for 4 weeks
  Interventions: Drug: olmesartan medoxomil oral tablets, hydrochlorothiazide oral tablets

INTERVENTIONS:
Other: placebo — Placebo oral tablets for 2 weeks
  Arms: 1
Drug: olmesartan medoxomil — olmesartan medoxomil oral tablets for 8 weeks
  Arms: 2
Drug: olmesartan medoxomil oral tablets, hydrochlorothiazide oral tablets — olmesartan medoxomil oral tablets,or olmesartan medoxomil oral tablets + hydrochlorothiazide oral tablets
  Arms: 3

SUMMARY:
To test the efficacy and safety of olmesartan in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 (19 if required by local authorities) to 75 years
* Males and females of any race. Female participants must take adequate contraceptive measures (oral contraceptives, I.U.D.), be post-menopausal or surgically sterilized
* Essential hypertension: sitting DBP greater than or equal to 90 and less than 110 mmHg
* Written Informed Consent
* Mentally competent
* Negative pregnancy test in women at a childbearing age at the beginning of the study

Exclusion Criteria:

* Patients with known severe (World Health Organization (WHO) stage III, sitting DBP stable at greater than or equal to 110 mmHg), malignant or secondary hypertension
* Patients who have had a myocardial infarction or percutaneous transluminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG) within the last 6 months
* Patients with a history or current evidence of congestive heart failure
* Bilateral renal artery stenosis
* Severe renal insufficiency (serum creatinine greater than 200 micro mol/l)
* Severe hepatic impairment or biliary obstruction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2333 (Actual)
Dates: Start 2002-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy on diastolic blood pressure of 40 mg olmesartan to a combination of 20 mg olmesartan and 12.5 mg hydrochlorothiazide in patients who are not sufficiently responding to treatment with 20 mg olmesartan. | From week 8 to week 12

SECONDARY OUTCOMES:
To assess the effects on systolic and diastolic blood pressure of 20 mg olmesartan, 40 mg olmesartan and the combination of 20 mg olmesartan with 12.5 mg hydrochlorothiazide at week 2, 4, 8 and 12. | 12 weeks
To detect less frequent adverse drug reactions and assess the safety and tolerability of olmesartan. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Michael Bohm, MD, Principal Investigator — Universitatskliniken des Saarlandes, Homburg, Germany
Locations (8):
- Result Cro, Vienna, Austria
- INPUT GmbG, Aachen, Germany
- Biokos Farma s.r.l., Bologna, Italy
- IMRO TRAMARKO International bv, Berghem, Netherlands
- EUROTRIALS Lda, Lisbon, Portugal
- Phidea S.L., Madrid, Spain
- PFC Pharma Focus Consultants AG, Zurich, Volketswil, Switzerland
- Inveresk Ltd., Edinburgh, United Kingdom